CLINICAL TRIAL: NCT01082991
Title: Strategies to Predict and Prevent In-Hospital Cardiac Arrest
Brief Title: Patient Acuity Rating: a Tool to Prevent In-Hospital Cardiac Arrest
Acronym: PAR
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15723A; 1K23HL097157-01 (NIH)
Record Dates: First submitted 2010-03-05; First posted 2010-03-09 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Heart Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prevention (Other)
  Interventions: Other: Preemptive Rapid Response Team intervention

INTERVENTIONS:
Other: Preemptive Rapid Response Team intervention — Non-ICU inpatients will be randomized on admission to an RRT surveillance group or standard of care. Daily risk prediction scores will be collected for all non-ICU inpatients. Those with high scores, who have been randomized to the surveillance arm, will be included on a list of patients, updated daily, that the Rapid Response Team will receive, with instructions to evaluate and intervene, if required, without waiting for formal activation by the usual channels.

SUMMARY:
The purpose of this study is to evaluate the accuracy of medical personnel in their ability to predict the likelihood of non-intensive care (ICU), ward patients to clinically deteriorate (defined as a cardiac arrest, unplanned ICU transfer, or unexpected death)via the use of a clinical judgement-based tool designed for this study, Patient Acuity Rating (PAR), to predict short-term clinical deterioration. We will compare the ability of this tool to predict clinical deterioration compared to accepted physiology-based tools and tools combining judgment and physiology as well as other markers of deterioration such as physician order changes. We will compare the sensitivity, specificity and area under the curve of these combined models to the predictive models including only physiology or clinical judgment. We will assess the correlation between specific physician orders and patient deterioration to determine whether specific clinical activities, such as emergently obtained radiology exams, predict impending deterioration. We hypothesize that PAR will be a useful tool for predicting clinical deterioration across the institution and that it will have a higher average accuracy for predicting clinical deterioration in non-ICU inpatients within 24 hours than the physiology-based tools alone. We further hypothesize that a combined metric which includes both the PAR and the individual physiologic components that comprise physiologic tools will not significantly improve prediction over the PAR alone. We further propose to use PAR to prospectively risk stratify patients for preemptive evaluation by the Rapid Response Team. We hypothesize that intervening on high risk patients by preemptively activating the hospital's Rapid Response Team (to assess and treat patients as needed) will decrease cardiac arrest rates and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Non-ICU ward inpatients
* PAR of 5 or above
* Ages 18+ years

Exclusion Criteria:

* ICU or outpatients
* PAR of 4 or lower
* Ages 17 years and under

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Mortality and cardiac arrest rates | 15 months
  Non-ICU ward inpatients will be randomized on admission to an RRT surveillance group or standard of care. Daily risk prediction scores will be collected for all non-ICU inpatients. Those with high scores, who have been randomized to the surveillance arm, will be included on a list of patients, updated daily, that the Rapid Response Team will receive, with instructions to evaluate and intervene, if required, without waiting for formal activation by the usual channels. Outcomes for these patients will be compared to those with comparable risk scores who were randomized to the control group.

SECONDARY OUTCOMES:
Length of stay | 15 months
Cost | 15 months
Time to ICU transfer | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Dana P Edelson, MD, MS, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Phillips AW, Yuen TC, Retzer E, Woodruff J, Arora V, Edelson DP. Supplementing cross-cover communication with the patient acuity rating. J Gen Intern Med. 2013 Mar;28(3):406-11. doi: 10.1007/s11606-012-2257-4. Epub 2012 Nov 6. PMID 23129163